CLINICAL TRIAL: NCT01442675
Title: Safety and Immunogenicity of a Single Dose of Menactra® Vaccine 4-6 Years After Prior Menactra Vaccine
Brief Title: Study of a Single Dose of Menactra® Vaccine 4-6 Years After Prior Menactra Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTA77; U1111-1117-7012 (Other: WHO)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection; Menactra®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meningococcal vaccine Group (Experimental): Participants must have received Menactra vaccine 4 to 6 years prior to enrollment
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate: Menactra®

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate: Menactra® — 0.5 mL, Intramuscular
  Other Names: Menactra®

SUMMARY:
The purpose of this trial is to describe the safety and antibody response to revaccination with Menactra vaccine in persons who received their first dose at ≥11 years of age.

Primary Objective:

- To evaluate the antibody responses to meningococcal serogroups A, C, Y, and W-135, measured by serum bactericidal assay using human complement (SBA-HC), induced by Menactra vaccine in subjects who were first vaccinated with Menactra 4-6 years ago.

Secondary Objective:

- To evaluate the antibody responses to serogroups A, C, Y, and W-135 in serum specimens collected 6 days post-vaccination in a subset of study population.

Observational Objective:

- To describe the rates of immediate reactions, solicited injection-site and systemic reactions, unsolicited adverse events and serious adverse events following vaccination.

DETAILED DESCRIPTION:
All participants will receive one dose of Menactra vaccine at their first clinic visit. There will be a telephone safety follow-up contact at six months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Received Menactra 4 to 6 years prior to enrollment, at an age ≥11 years, and is < 56 years of age on the day of enrollment.
* Informed consent form has been signed and dated by the subject or by the subject and the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of child bearing potential without using an effective method of contraception or not practicing abstinence for at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. Females who are pre-menarche or post-menopausal for at least 1 year, or surgically sterile will not be excluded.
* Any condition which, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* History of documented invasive meningococcal disease.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study.
* Suspected or known hypersensitivity to latex or to any of the components of Menactra vaccine, or history of a life-threatening reaction to Menactra vaccine or to a vaccine containing any of the same substances.
* Receipt of any meningococcal vaccine since receipt of a single dose of Menactra vaccine 4-6 years prior to enrollment.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before the Day 28 visit; except that influenza vaccine may have been received between 30 and 15 days (but no less than 15 days) before receiving study vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of laboratory-confirmed seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, as reported by the subject.
* Personal history of Guillain-Barré syndrome (GBS).
* Laboratory-confirmed thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug use that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Receipt of oral or injectable antibiotic therapy within the 72 hours prior to the first blood draw.
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective subject should not be enrolled in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 834 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (15):
- United States (15):
  - Little Rock, Arkansas
  - San Diego, California
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Spokane, Massachusetts
  - Woburn, Massachusetts
  - Niles, Michigan
  - Stevensville, Michigan
  - Rochester, New York
  - Cleveland, Ohio
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Layton, Utah
  - Orem, Utah
  - Midlothian, Virginia

REFERENCES:
- [Derived] Robertson CA, Greenberg DP, Hedrick J, Pichichero M, Decker MD, Saunders M. Safety and immunogenicity of a booster dose of meningococcal (groups A, C, W, and Y) polysaccharide diphtheria toxoid conjugate vaccine. Vaccine. 2016 Oct 17;34(44):5273-5278. doi: 10.1016/j.vaccine.2016.09.003. Epub 2016 Sep 15. PMID 27642132
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 26 September 2011 through 21 December 2011 at 15 clinic centers in the United States.
Pre-assignment Details: A total of 834 participants who met all of the inclusion and none of the exclusion criteria were randomized; 831 were vaccinated in this study.
Groups:
- Menactra® Vaccine Group: Participants <56 years of age who received Menactra vaccine 4-6 years previously at age ≥11 years received a single dose of Menactra vaccine in this study.
Period: Overall Study
Arm/Group | Menactra® Vaccine Group
Started | 834
Safety Analysis Set | 831 (Safety Analysis Set are subjects who received study vaccine and for whom safety data were available.)
Per-Protocol Analysis Set | 781 (The Per-Protocol Analysis Set are subjects with no pre-defined protocol deviations.)
Completed | 822
Not Completed | 12
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Menactra® Vaccine Group: Participants <56 years of age who received Menactra vaccine 4-6 years previously at age ≥11 years received a single dose of Menactra in this study.
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 834
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 592
  Between 18 and 65 years | 242
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 17.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 434
  Male | 400
Region of Enrollment [Number; unit: Participants]
  United States | 834

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Antibody Titers ≥1:8 Against Meningococcal Serogroups A, C, Y, and W-135 by Serum Bactericidal Assay Using Human Complement Following Vaccination With Menactra®
Description: Meningococcal antibodies against serogroups A, C, Y, and W-135 were assessed by serum bactericidal assay using human complement (SBA-HC)
Time Frame: Day 28 post-vaccination
Population: SBA-HC antibody titers were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Participants
  Serogroup A | 776
  Serogroup C | 778
  Serogroup Y | 779
  Serogroup W-135 | 780

2. Secondary Outcome: Number of Participants Achieving Antibody Titers ≥1:4 Against Meningococcal Serogroups A, C, Y, and W-135 by Serum Bactericidal Assay Using Human Complement Before and Following Vaccination With Menactra®
Description: Meningococcal antibodies against serogroups A, C, Y, and W-135 were assessed by serum bactericidal assay using human complement (SBA-HC).
  Serum samples were collected from a random subset of vaccinated participants 6 days post-vaccination to assess SBA-HC antibody titers at this time point.
Time Frame: Day 0 (pre-vaccination), Day 6 and Day 28 post-vaccination
Population: SBA-HC antibody titers were assessed in the Per-protocol Analysis Set. Serum samples were collected from a random subset of vaccinated participants 6 days post-vaccination to assess SBA-HC antibody titers at this time point.
Measure: Number; unit: Participants
Groups:
- Menactra® Vaccine Group: Participants <56 years of age who received Menactra 4-6 years previously at age ≥11 years received a single dose of Menactra vaccine
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Participants
  Serogroup A (Day 0 pre-vaccination; N=781) | 675
  Serogroup A (Day 6 post-vaccination; N=112) | 110
  Serogroup A (Day 28 post-vaccination; N=781) | 781
  Serogroup C (Day 0 pre-vaccination; N=781) | 443
  Serogroup C (Day 6 post-vaccination; N=112) | 112
  Serogroup C (Day 28 post-vaccination; N=781) | 780
  Serogroup Y (Day 0 pre-vaccination; N=781) | 389
  Serogroup Y (Day 6 post-vaccination; N=112) | 111
  Serogroup Y (Day 28 post-vaccination; N=781) | 780
  Serogroup W-135 (Day 0 pre-vaccination; N=781) | 604
  Serogroup W-135 (Day 6 post-vaccination; N=112) | 111
  Serogroup W-135 (Day 28 post-vaccination; N=781) | 780

3. Secondary Outcome: Number of Participants Achieving Antibody Titers ≥1:8 Against Meningococcal Serogroups A, C, Y, and W-135 by Serum Bactericidal Assay Using Human Complement Before and Following Vaccination With Menactra®
Description: as for outcome 2
Time Frame: Day 0 (pre-vaccination), Day 6 and Day 28 post-vaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Participants
  Serogroup A (Day 0 pre-vaccination; N=781) | 504
  Serogroup A (Day 6 post-vaccination; N=112) | 110
  Serogroup A (Day 28 post-vaccination; N=781) | 776
  Serogroup C (Day 0 pre-vaccination; N=781) | 345
  Serogroup C (Day 6 post-vaccination; N=112) | 111
  Serogroup C (Day 28 post-vaccination; N=781) | 778
  Serogroup Y (Day 0 pre-vaccination; N=781) | 302
  Serogroup Y (Day 6 post-vaccination; N=112) | 111
  Serogroup Y (Day 28 post-vaccination; N=781) | 779
  Serogroup W-135 (Day 0 pre-vaccination; N=781) | 535
  Serogroup W-135 (Day 6 post-vaccination; N=112) | 111
  Serogroup W-135 (Day 28 post-vaccination; N=781) | 780

4. Secondary Outcome: Number of Participants Achieving At Least Four-Fold Rise in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers by Serum Bactericidal Assay Using Human Complement Following Vaccination With Menactra®
Description: as for outcome 2
Time Frame: Day 6 and Day 28 post-vaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Participants
  Serogroup A (Day 6 post-vaccination; N=112) | 97
  Serogroup A (Day 28 post-vaccination; N=781) | 742
  Serogroup C (Day 6 post-vaccination; N=112) | 102
  Serogroup C (Day 28 post-vaccination; N=781) | 744
  Serogroup Y (Day 6 post-vaccination; N=112) | 106
  Serogroup Y (Day 28 post-vaccination; N=781) | 758
  Serogroup W-135 (Day 6 post-vaccination; N=112) | 103
  Serogroup W-135 (Day 28 post-vaccination; N=781) | 750

5. Secondary Outcome: Geometric Mean Antibody Titers Against Meningococcal Serogroups A, C, Y, and W-135 by Serum Bactericidal Assay Using Human Complement Before and Following Vaccination With Menactra®
Description: as for outcome 2
Time Frame: Day 0 (pre-vaccination), Day 6 and Day 28 post-vaccination
Population: Geometric mean titers (GMTs) were assessed in the Per-protocol Analysis Set. Serum samples were collected from a random subset of vaccinated participants 6 days post-vaccination to assess SBA-HC GMTs at this time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Titers
  Serogroup A (Day 0 pre-vaccination; N=781) | 8.9 [8.3 to 9.6]
  Serogroup A (Day 6 post-vaccination; N=112) | 227.6 [166.4 to 311.3]
  Serogroup A (Day 28 post-vaccination; N=781) | 421.2 [378.8 to 468.3]
  Serogroup C (Day 0 pre-vaccination; N=781) | 8.8 [7.8 to 10.0]
  Serogroup C (Day 6 post-vaccination; N=112) | 639.8 [457.4 to 895.0]
  Serogroup C (Day 28 post-vaccination; N=781) | 1135 [1013.0 to 1271.8]
  Serogroup Y (Day 0 pre-vaccination; N=781) | 6.2 [5.6 to 6.9]
  Serogroup Y (Day 6 post-vaccination; N=112) | 655.8 [474.8 to 905.9]
  Serogroup Y (Day 28 post-vaccination; N=781) | 1303.6 [1183.1 to 1436.4]
  Serogroup W-135 (Day 0 pre-vaccination; N=781) | 13.8 [12.4 to 15.3]
  Serogroup W-135 (Day 6 post-vaccination; N=112) | 702 [508.0 to 970.2]
  Serogroup W-135 (Day 28 post-vaccination; N=781) | 1271.6 [1145.3 to 1411.8]

6. Secondary Outcome: Geometric Mean Antibody Titer Ratios Against Meningococcal Serogroups A, C, Y, and W-135 by Serum Bactericidal Assay Using Human Complement Following Vaccination With Menactra®
Description: as for outcome 2
Time Frame: Day 6 and Day 28 post-vaccination
Population: Geometric mean titers ratios (GMTRs) were assessed in the Per-protocol Analysis Set. Serum samples were also collected from a random subset of vaccinated participants 6 days post-vaccination to assess SBA-HC GMTRs at this time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers ratio
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 781
Titers ratio
  Serogroup A (Day 6 post-vaccination; N=112) | 30.5 [21.8 to 42.5]
  Serogroup A (Day 28 post-vaccination; N=781) | 47.2 [42.3 to 52.7]
  Serogroup C (Day 6 post-vaccination; N=112) | 64 [42.7 to 95.9]
  Serogroup C (Day 28 post-vaccination; N=781) | 128.3 [112.0 to 147.0]
  Serogroup Y (Day 6 post-vaccination; N=112) | 121.1 [84.5 to 173.5]
  Serogroup Y (Day 28 post-vaccination; N=781) | 209.1 [184.4 to 237.1]
  Serogroup W-135 (Day 6 post-vaccination; N=112) | 45.5 [31.0 to 67.0]
  Serogroup W-135 (Day 28 post-vaccination; N=781) | 92.4 [81.1 to 105.4]

7. Secondary Outcome: Number of Participants Reporting Solicited Injection-Site or Systemic Reactions Following Vaccination With Menactra®
Description: Solicited injection-site reactions: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering. Grade 3 injection-site reactions: Pain - Significant, prevents daily activity; Erythema and Swelling - >100 mm. Grade 3 systemic reactions: Fever - ≥40˚C or ≥104˚F; Headache, Malaise, Myalgia, and Shivering - Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 831
Participants
  Injection-site Pain (N=821) | 494
  Grade 3 Injection-site Pain (N=821) | 20
  Injection-site Erythema (N=821) | 10
  Grade 3 Injection-site Erythema (N=821) | 0
  Injection-site Swelling (N=821) | 14
  Grade 3 Injection-site Swelling (N=821) | 0
  Fever (N=817) | 6
  Grade 3 Fever (N=817) | 0
  Headache (N=822) | 317
  Grade 3 Headache (N=822) | 22
  Malaise (N=822) | 242
  Grade 3 Malaise (N=822) | 23
  Myalgia (N=822) | 352
  Grade 3 Myalgia (N=822) | 19
  Shivering (N=822) | 102
  Grade 3 Shivering (N=822) | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 6 months post-vaccination.
Description: The solicited injection site and systemic reactions were recorded in a diary card within 7 days of vaccination; the total number (N) reflects those subjects for which the diary cards were returned and for which data were available for the event during the period.
Groups:
- Menactra® Vaccine Group: Participants <56 years of age who received Menactra 4-6 years previously at age >= 11 years received a single dose of Menactra vaccine
Arm/Group | Menactra® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 11/831
Other Adverse Events (participants affected / at risk) | 494/831
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Vaccine Group (N=831)
Bronchitis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menactra® Vaccine Group (N=831)
Injection site Pain (General disorders) | 494/821 (494)
Headache (Nervous system disorders) | 317/822 (317)
Malaise (General disorders) | 242/822 (242)
Myalgia (Musculoskeletal and connective tissue disorders) | 352/822 (352)
Shivering (General disorders) | 102/822 (102)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications